CLINICAL TRIAL: NCT04791137
Title: Feasibility Randomized Controlled Trial Using a 'Leapfrog' Design: Optimizing an Internet-delivered Cognitive Training Intervention to Reduce Anhedonia
Brief Title: Feasibility Randomized Controlled Trial Using a 'Leapfrog' Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Simon Blackwell, Postdoctoral Researcher, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 365
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Anhedonia; Depression
Keywords: Cognitive Bias Modification; Mental Imagery; Leapfrog Design
MeSH Terms: conditions — Anhedonia; Depression

STUDY DESIGN:
Intervention Model Description: The leapfrog trial design is a parallel-arm design in which participants and randomly allocated to one of several treatment arms on a 1:1:1... ratio. One trial arm is designated the comparison arm, and all other arms are compared to this comparison arm via sequential Bayesian analyses. Depending on the outcomes of the sequential analyses (based on reaching Bayes Factor thresholds for 'success' or 'failure', trial arms may be removed, or take the place of the comparison arm while the trial is ongoing, and new arms may also be introduced into an ongoing trial.
Who Masked: Participant
Masking Description: Participants are not blind as to whether they are receiving an intervention or monitoring only, but otherwise are blind to the status of which intervention they are receiving, i.e. 'original' version of the imagery CBM or an attempted improvement. Researchers are not blind to participant allocations, but the study is planned to be mostly automated, reducing opportunities to influence participants. Researchers will monitor performance of the arms as data accumulates, via the sequential analyses, and will therefore not be blind to outcomes as the trial progresses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Monitoring (No Intervention): Participants complete weekly questionnaires (QIDS-SR, PMH, GAD-7) on a weekly basis but receive no intervention.
- Standard imagery cognitive bias modification (Experimental): Participants are scheduled to complete a first introductory session then 12 further training sessions of a 'standard' imagery cognitive bias modification (CBM) intervention derived from that implemented in previous studies.
  Interventions: Behavioral: Imagery cognitive bias modification
- Standard imagery cognitive bias modification plus additional rationale and transfer instructions (Experimental): Participants are scheduled to complete a first introductory session then 12 further training sessions of a 'standard' imagery cognitive bias modification (CBM) intervention, but in addition are first presented with a more extended rationale for completing the training, and during each training session are provided with instructions to practice retrieval and rehearsal of the training contents in between sessions.
  Interventions: Behavioral: Imagery cognitive bias modification
- Standard imagery cognitive bias modification with frequent brief sessions (Experimental): Participants are scheduled to complete a first introductory session then 40 brief (~5 min) sessions of a 'standard' imagery cognitive bias modification (CBM) intervention, with 2 per day five days per week for each of the four training weeks. In addition, as with the arm "Standard imagery cognitive bias modification plus additional rationale and transfer instructions", participants are first presented with a more extended rationale for completing the training, and during many of the training sessions are provided with instructions to practice retrieval and rehearsal of the training contents in between sessions. This arm was added into the ongoing trial on 30.05.21.
  Interventions: Behavioral: Imagery cognitive bias modification
- Standard imagery cognitive bias modification with a less intensive schedule (Experimental): Participants are scheduled to complete a first introductory session then 11 further sessions of a 'standard' imagery cognitive bias modification (CBM) intervention, with 3 sessions scheduled for each of the four training weeks. Sessions have fewer training scenarios than the "Standard imagery cognitive bias modification" condition and more varied task instructions. In addition, as with the arm "Standard imagery cognitive bias modification plus additional rationale and transfer instructions", participants are first presented with a more extended rationale for completing the training, and during many of the training sessions are provided with instructions to practice retrieval and rehearsal of the training contents in between sessions. This arm was added into the ongoing trial on 09.06.21.
  Interventions: Behavioral: Imagery cognitive bias modification

INTERVENTIONS:
Behavioral: Imagery cognitive bias modification — The imagery cognitive bias modification intervention is derived from that developed via experimental psychopathology research (e.g. Holmes et al., 2009) and adapted for clinical applications in the context of depression (e.g. Blackwell & Holmes, 2010; Blackwell et al., 2015). The intervention is a series of training sessions in which participants listen to training scenarios consisting of descriptions of everyday situations, structured so that they start ambiguously but always end positively. Participants are instructed to imagine themselves in the situations described as the scenarios unfold. It is hypothesised that via repeatedly practising imagining positive resolutions for ambiguous situations in the training sessions, a bias is trained to automatically imagine positive resolutions for ambiguous situations encountered in daily life.
  Arms: Standard imagery cognitive bias modification; Standard imagery cognitive bias modification plus additional rationale and transfer instructions; Standard imagery cognitive bias modification with a less intensive schedule; Standard imagery cognitive bias modification with frequent brief sessions

SUMMARY:
This study is a small-scale randomized controlled trial (RCT) using a 'Leapfrog' design (Blackwell, Woud, Margraf, & Schönbrodt, 2019) with the aim of investigating feasibility of this design in the context of an RCT of an internet-delivered intervention. The leapfrog design will be applied to a simple cognitive training intervention, imagery cognitive bias modification (imagery CBM), completed over a four-week training period. The trial will start with the three arms described in the initial registration, but these will be removed and new arms added over the course of the trial on the basis of sequential Bayesian analyses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Fluent German
* Willing and able to complete all study procedures (including having a suitable device/ internet access)
* Interested in monitoring their mood over the study time-period (one month)
* Score of ≥ 6 on the Quick Inventory of Depressive Symptomatology, including ≥ 1 on item 13 (General Interest), indicating at least mild levels of depression symptoms and anhedonia

Exclusion Criteria:

* No exclusion criteria set

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Dimensional Anhedonia Rating Scale (DARS) | Post-intervention (4 weeks post-baseline).
  A 17-item scale measuring anhedonia (Rizvi et al., 2015). The primary analysis is a between-groups comparison of post-intervention scores, controlling for baseline scores, using constrained longitudinal data analysis (cLDA). An approximate Bayes factor is then calculated via the t-statistic for the Time x Group effect with a directional default Cauchy prior (rscale parameter = √2/2).

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report (QIDS) | Baseline, 1 week post-baseline, 2 weeks post-baseline, 3 weeks post-baseline, post-intervention (4 weeks post-baseline)
  A 15-item version of the QIDS (Rush et al., 2013), excluding the suicidal ideation item, will be used
GAD-7 | Baseline, 1 week post-baseline, 2 weeks post-baseline, 3 weeks post-baseline, post-intervention (4 weeks post-baseline)
  A brief 7-item measure of generalized anxiety symptoms (Spitzer et al., 2006)
Positive Mental Health Scale (PMH) | Baseline, 1 week post-baseline, 2 weeks post-baseline, 3 weeks post-baseline, post-intervention (4 weeks post-baseline)
  A 9-item questionnaire designed to assess positive mental health (Lukat et al., 2016)
Ambiguous Scenarios Test for Depression (AST) | Baseline and post-intervention (4 weeks post-baseline)
  A measure with two 15-item parallel forms designed to assess depression-relevant negative interpretation biases (Rochbacher & Reinecke, 2014)
Prospective Imagery Test (PIT) | Baseline and post-intervention (4 weeks post-baseline)
  A measure designed to assess vividness of positive and negative future-oriented imagery (Stöber et al., 2000), here administered with as two 10-item parallel versions (each with 5 positive and 5 negative items).
Negative Effects Questionnaire - Short Form (NEQ) | Post-intervention (4 weeks post-baseline)
  A 20-item questionnaire designed to assess potential negative effects of psychological interventions (Rozental et al., 2019)

OTHER OUTCOMES:
Spontaneous Use of Imagery Scale (SUIS) | Baseline
  A 12-item questionnaire assessing experience of spontaneous non-emotional mental imagery in daily life (Reisberg et al., 2003)
Credibility / Expectancy Questionnaire (CEQ) | Baseline
  A 6-item questionnaire assessing participants' evaluation of the credibility of an intervention (3 items) and their expectancy of symptom improvement (3 items) over the course of an intervention (Devilly & Borkovec, 2000)
Feedback questionnaire | Post-intervention (4 weeks post-baseline)
  A questionnaire containing both rating scales and open questions for eliciting participants' feedback about the study and interventions completed (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Simon E Blackwell, Dr. phil., Principal Investigator — Ruhr-Universität Bochum
Locations (1):
- Ruhr University of Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on publication via a suitable repository such as the Open Science Framework, and will be made available to reviewers at the time of submission (or publically with a pre-print version of the manuscript). Data made available will be the research data reported in the publication, with the exception of any data that could compromise participant anonymity.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Supporting information will be made available on publication via a suitable repository such as the Open Science Framework, and will be made available to reviewers at the time of submission (or publically with a pre-print version of the manuscript).
URL: https://osf.io/8mxda/

REFERENCES:
- [Background] Blackwell, S. E., Woud, M. L., Margraf, J., & Schönbrodt, F. D. (2019). Introducing the leapfrog design: A simple Bayesian adaptive rolling trial design for accelerated treatment development and optimization. Clinical Psychological Science, 7, 1222-1243. https://doi.org/10.1177/2167702619858071
- [Derived] Blackwell SE, Schonbrodt FD, Woud ML, Wannemuller A, Bektas B, Braun Rodrigues M, Hirdes J, Stumpp M, Margraf J. Demonstration of a 'leapfrog' randomized controlled trial as a method to accelerate the development and optimization of psychological interventions. Psychol Med. 2023 Oct;53(13):6113-6123. doi: 10.1017/S0033291722003294. Epub 2022 Nov 4. PMID 36330836
- See also: Link for participants to enrol — https://homepage.ruhr-uni-bochum.de/Simon.Blackwell/mio-studie.html?st=lf3&so=c0